CLINICAL TRIAL: NCT04810702
Title: Impact of Von Willebrand Factor and Its Multimers on Angiogenesis
Acronym: WILLANGIO
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0531
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — frozen plasma fractions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with von Willebrand disease
  Interventions: Other: no intervention
- case control
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The study aims to study the expression of numerous proteins involved in angiogenesis in 70 patients with von Willebrand disease in order to try to identify markers of interest. Secondly, the investigators plan to investigate whether there is a relationship between the proteins tested, the distribution of multimers and the clinical phenotype of the patients, in particular by looking for the presence of bleeding linked to the presence of angiodysplasias.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patient with von Willebrand disease proven by genetic analysis of the VWF gene.
* Lack of treatment that could interfere with angiogenesis.
* Patient informed by an information note sent to his home, with the possibility of objecting to the use of his blood samples in the context of research.

For the control:

* Patient with a normal coagulation report
* Absence of abnormal hemorrhagic symptoms
* Lack of notion of angiodysplasia.
* Lack of treatment that could interfere with angiogenesis.
* Patient informed by an information note sent to his home, with the possibility of objecting to the use of his blood samples in the context of research.

Exclusion Criteria:

* Patient under guardianship or curatorship.
* Pregnant and lactating women.
* Blood transfusion or treatment with von Willebrand factor concentrates less than 7 days old.
* Treatment which may interfere with angiogenesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The studied population will be composed of:
  * 70 patients with von Willebrand disease: 10 type 1 patients, 10 type 2A (IIA) patients, 10 type 2A (IIE) patients, 10 type 2B patients, 10 type 2M patients, 10 type 2M patients (2A-like) and 10 type 3 patients.
  * 20 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-08-07 (Estimated)

PRIMARY OUTCOMES:
To study the relationship between proteins involved in angiogenesis and the distribution of multimers in patients with von Willebrand disease in order to define markers of interest | 1 year
  Compare the distribution of multimers assays between different groups of patients and the control group
To study the relationship between proteins involved in angiogenesis and the distribution of multimers in patients with von Willebrand disease in order to define markers of interest | 1 year
  Compare the distribution of protein assays between different groups of patients and the control group

SECONDARY OUTCOMES:
To study the relationship between the distribution of multimers and the clinical phenotype of patients, and in particular the presence of angiodysplasias | 1 year
  To study the correlation between the clinical phenotype and the assays of angiogenesis proteins
To study the relationship between the markers of interest and the clinical phenotype of patients, and in particular the presence of angiodysplasias | 1 year
  To study the correlation between the clinical phenotype and the distribution of multimers

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided